CLINICAL TRIAL: NCT03294408
Title: Capacity of Multimodal Imaging of Subchondral Bone for the Prediction of Structural Evolution in Knee Osteoarthritis
Brief Title: Multimodal Imaging of Subchondral Bone in Knee Osteoarthritis : Predictive Model
Acronym: MOSART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: University of Nancy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2016-01; 2016-A00552-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2017-07-04; First posted 2017-09-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Joint Disease; Arthritis; Musculoskeletal Disease
Keywords: fractal analysis; trabecular bone texture; knee osteoarthritis; subchondral bone; Medical Resonnance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthritis; Musculoskeletal Diseases | interventions — Multimodal Imaging

STUDY DESIGN:
Intervention Model Description: Interventional study among patients suffering from knee osteoarthritis for at least six months. All the patients will benefit from a multimodal imaging and clinical assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging (Other): multimodal imaging and clinical assessment
  Interventions: Diagnostic Test: multimodal imaging

INTERVENTIONS:
Diagnostic Test: multimodal imaging
  Other Names: clinical assessment

SUMMARY:
Predictive factors of osteoarthritis progression are not yet well understood. However, a growing role attaches importance to the subchondral bone. The aim of the present project is to determine predictive factors of progression of osteoarthritis at the knee by a multimodal characterization of subchondral bone by Medical Resonnance Imaging, direct high resolution digitization radiographs and bone texture analysis. At the end of the project, an innovative imaging device, combining semi-automatic softwares for texture analysis, control detection and image registration would be supplied. This will enable on the one hand a more accurate and reproducible way to measure the joint space width of the affected compartment and on the other hand, an assistance to better detect patients at risk of progression of their knee osteoarthritis. Identifying These "progressors" patients might permit their selection in clinical trials at baseline adapted to their severe disease, using for example biologic treatments targeting knee osteoarthritis. The main objective of this study is to analyze the predictive capacities of bone texture parameters measured on the high-resolution radiography of the knee on the structural evolution of the knee osteoarthritis at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis according to the criteria of knee osteoarthritis of American College of Rheumatology.
* Having felt a painful push in the last 6 months.
* Visual Analogic Scale pain > 4 on a 0 to 10 scale.
* having a Radiographic score of OARSI (Osteoarthritis Research Society International Score) from 2 to 3 whether it is for the presence of a joint space narrowing or the presence of an osteophyte

Exclusion Criteria:

* Patello-femoral degenerative osteoarthritis isolated.
* Incapacitated to consider the position in schuss for the realization of the radiography.
* Valgus > in 5 °
* Secondary degenerative osteoarthritis

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have one-point increase in the quality score of OARSI | 3 years
  Patients who over the 3-year follow-up period will have a one-point increase in the quality score of OARSI compared to the initial pinch score (Altman RD et al, Osteoarthritis and Cartilage 1995).
Proportion of patients whose joint space reduction is greater than the smallest reliable detectable difference. | 3 years
  Patients whose joint space reduction is greater than the smallest reliable detectable difference.
Proportion of patients who have a decrease in joint space of 0.5 mm | 3 years
  Patients who have a decrease in joint space of 0.5 mm or more over the 3-year period (Cooper C et al, CMRO 2012).

SECONDARY OUTCOMES:
Proportion of patients who have evolution of medial femoral tibial joint space | 3 years
  Evolution of medial femoral-tibial joint space
Number of particpants who will have evolution of strucutral lesion score | 3 years
  Evolution structural lesion score is OARSI (OsteoArthritis Research Society International score)
Evolution of algo-functional scores (OAKHQOL) | 3 years
  OAKHQOL (OsteoArthritis of Knee and Hip Quality Of Life) scores
Evolution of algo-functional scores (WOMAC) | 3 years
  WOMAC (McMaster Western Ontario questionnaire ) scores
Change From Baseline in quality of life Scores | 3 years
  Short Form 36
Change From Baseline in Pain Scores on the Visual Analog Scale | 3 years
  Pain visual analogical score

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, Dr, Principal Investigator — CHR Orléans
Locations (2):
- France (2):
  - Chu Brabois, Nancy
  - CHR Orléans, Orléans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janvier T, Jennane R, Valery A, Harrar K, Delplanque M, Lelong C, Loeuille D, Toumi H, Lespessailles E. Subchondral tibial bone texture analysis predicts knee osteoarthritis progression: data from the Osteoarthritis Initiative: Tibial bone texture & knee OA progression. Osteoarthritis Cartilage. 2017 Feb;25(2):259-266. doi: 10.1016/j.joca.2016.10.005. Epub 2016 Oct 11. PMID 27742531
- [Background] Arden N, Richette P, Cooper C, Bruyere O, Abadie E, Branco J, Brandi ML, Berenbaum F, Clerc C, Dennison E, Devogelaer JP, Hochberg M, D'Hooghe P, Herrero-Beaumont G, Kanis JA, Laslop A, Leblanc V, Maggi S, Mautone G, Pelletier JP, Petit-Dop F, Reiter-Niesert S, Rizzoli R, Rovati L, Tajana Messi E, Tsouderos Y, Martel-Pelletier J, Reginster JY. Can We Identify Patients with High Risk of Osteoarthritis Progression Who Will Respond to Treatment? A Focus on Biomarkers and Frailty. Drugs Aging. 2015 Jul;32(7):525-35. doi: 10.1007/s40266-015-0276-7. PMID 26085027
- [Background] Woloszynski T, Podsiadlo P, Stachowiak GW, Kurzynski M, Lohmander LS, Englund M. Prediction of progression of radiographic knee osteoarthritis using tibial trabecular bone texture. Arthritis Rheum. 2012 Mar;64(3):688-95. doi: 10.1002/art.33410. PMID 21989629
- [Background] Guermazi A, Roemer FW, Felson DT, Brandt KD. Motion for debate: osteoarthritis clinical trials have not identified efficacious therapies because traditional imaging outcome measures are inadequate. Arthritis Rheum. 2013 Nov;65(11):2748-58. doi: 10.1002/art.38086. No abstract available. PMID 23861096
- [Background] Kraus VB, Feng S, Wang S, White S, Ainslie M, Brett A, Holmes A, Charles HC. Trabecular morphometry by fractal signature analysis is a novel marker of osteoarthritis progression. Arthritis Rheum. 2009 Dec;60(12):3711-22. doi: 10.1002/art.25012. PMID 19950282